CLINICAL TRIAL: NCT02053701
Title: Technical Developments for High-field Brain Magnetic Resonance Spectroscopy
Brief Title: High-field Brain Magnetic Resonance Spectroscopy
Status: Active, not recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1210M23141; P41EB015894 (NIH)
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: magnetic resonance spectroscopy; quantification precision; brain; brain metabolites

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Magnetic resonance spectroscopy (MRS) allows non-invasive measurement of the concentration of up to 18 metabolites in the brain ("neurochemical profile").

The objective of this proposal is to develop new methods for high-field brain MRS (3 to 7 Tesla).

Our main hypothesis is that higher magnetic fields lead to improved spatial and temporal resolution and improved quantification precision.

Aims

1. To obtain improved "neurochemical profiles" in the brain using single voxel proton MRS at very high field (3 Tesla to 7 Tesla).
2. To develop new methods for proton magnetic resonance spectroscopic imaging (MRSI) to obtain metabolic maps at very high field (3 Tesla to 7 Tesla).

Since this project is focused on technical development, only healthy volunteers will be recruited (no patients).

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old

Exclusion Criteria:

* no metallic implant or other MRI-incompatible device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-06-01 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Precision of quantification of brain metabolites concentrations | One time only
  This protocol is devoted exclusively to technical development and testing of MRS methods on our MR scanners. As such, there is no well-defined outcome measure or time frame. It is a continuous effort. We recruit subjects on an ongoing basis to test, optimize, and assess the performance of newly developed techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Gilles Henry, PhD, Principal Investigator — Center for Magnetic Resonance Research, University of Minnesota
Locations (1):
- Center for Magnetic Resonance Research, Minneapolis, Minnesota, United States